CLINICAL TRIAL: NCT02562573
Title: A Phase 2, Single-Arm, Open-Label Study to Evaluate the Safety and Tolerability of PBI-4050 in Type 2 Diabetes Patients With Metabolic Syndrome
Brief Title: Study to Evaluate the Safety and Tolerability of PBI-4050 in Type 2 Diabetes Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Liminal BioSciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBI4050-ATX-9-04
Record Dates: First submitted 2015-08-28; First posted 2015-09-29 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2016-10

CONDITIONS: Type 2 Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome | interventions — setogepram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PBI4050 (Experimental): Four 200 mg capsules (total 800 mg) administered orally, once a day.
  Interventions: Drug: PBI4050

INTERVENTIONS:
Drug: PBI4050

SUMMARY:
This is a Phase 2, open-label, single-arm study of the safety and tolerability of PBI-4050 800 mg daily oral administration in type 2 diabetes patients with metabolic syndrome.

A total of 12 patients will initially be enrolled for study participation. A Data Safety Monitoring Board (DSMB) will continuously review data obtained from the 12 patients. When the 12 patients have completed at least one month of study treatment, the DSMB will meet and determine whether additional patients may be enrolled or the study should be stopped. If the safety is deemed acceptable to continue with the study, the study will enroll a maximum of 36 patients.

DETAILED DESCRIPTION:
This Phase 2 study will be performed by 1 site in Canada. The total duration of study participation for each patient is at least 18 weeks and comprises 6 study visits.

Patients who choose to participate in the extension study will be in the study for a total of up to 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years of age or older.
2. Patient has signed written informed consent.
3. Patient has a clinical diagnosis of type 2 diabetes mellitus with a hemoglobin A1c (HbA1c) level between 7% and 10%.
4. Patient has been receiving stable antidiabetic therapy (oral agents with or without basal insulin given once daily in the evening) for a minimum of 3 months before the screening visit.
5. Patient is able and willing to self-monitor blood glucose level at home.
6. Patient has a body mass index (BMI) of at least 27 kg/m2.
7. Patient has metabolic syndrome, having at least 3 of the 5 metabolic syndrome risk factors.

Exclusion Criteria:

1. Patient requires intensive insulin therapy (defined as more than basal insulin given once daily in the evening) in addition to oral hypoglycemic agents for blood glucose control.
2. Patient has recent or on-going infection requiring systemic treatment with an anti-infective agent within 30 days before screening.
3. Patient has had at least one episode of severe hypoglycemia in the past 12 months, defined as having a blood glucose level < 3.0 mmol/L and/or requiring third party assistance to treat hypoglycemic episode.
4. Patient has evidence of significant cardiovascular disease, including myocardial infarction, unstable angina, coronary bypass surgery, percutaneous transluminal coronary angioplasty (PTCA), congestive heart failure (New York Heart Association Class III-IV), stroke, or severe ischemic disease within 3 months before screening.
5. Patient has uncontrolled hypertension with BP > 150/95 mm Hg.
6. Patient has a diagnosis of rheumatic or inflammatory disease, such as rheumatoid arthritis (RA), polymyalgia rheumatic (PMR), inflammatory bowel disease (IBD); or other autoimmune or inflammatory disease such as systemic lupus erythematosus (SLE) or psoriasis.
7. Patient is concurrently taking and plans to routinely continue taking anti-inflammatory medications, such as nonsteroidal anti-inflammatory drugs (NSAIDs) and corticosteroids, during the study.
8. Patient is currently using weight loss medications.
9. Patient has significantly elevated liver enzyme levels, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.5 × upper limit of normal (ULN) or total bilirubin above ULN.
10. Patient has a history of chronic alcohol or other substance abuse.
11. Woman who is pregnant, breast-feeding, or planning a pregnancy during the course of the study.
12. Woman of childbearing potential who is unwilling to use adequate birth control throughout the duration of the study.
13. Patient has any condition that, in the investigator's opinion, is likely to interfere with study conduct and compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal laboratory values and/or adverse events that are related to treatment | 7 months

SECONDARY OUTCOMES:
Change from baseline on waist circumference | 6 months
Change from baseline on biomarkers | 6 months
  % reduction and/or increase of biomarkers
Change from baseline on antidiabetic treatment | 6 months
  Treatment discontinued, dosing change, and/or new medication added
Change from baseline on triglycerides | 6 months
Change from baseline on BP | 6 months
Change from baseline on HDL-C | 6 Months
Change from baseline on fasting plasma glucose | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Edmonton, Alberta, Canada